CLINICAL TRIAL: NCT05542303
Title: A Single Ascending Dose, Safety, and Pharmacokinetic Study of ZB001 in Healthy Chinese Subjects
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of ZB001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZB001-01-001
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZB001 for injection (Experimental): Treated different dose cohorts with single intravenous injection of ZB001
  Interventions: Drug: ZB001 for injection

INTERVENTIONS:
Drug: ZB001 for injection — Dose Cohort1 (3mg/kg) ZB001 of single IV injection
Drug: ZB001 for injection — Dose Cohort2 (10mg/kg) ZB001 of single IV injection
Drug: ZB001 for injection — Dose Cohort3 (20mg/kg) ZB001 of single IV injection

SUMMARY:
The investigational drug, ZB001 is a humanized IgG1κ monoclonal antibody (mAb) targeting human IGF-1R. This clinical trial will examine the safety, tolerability, and pharmacokinetics (PK) of single ascending doses of ZB001 in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese subjects between 18 and 55 years old (inclusive) at Screening
2. Free of any clinically significant disease or medical condition at screening as determinedby the Investigator
3. Body weight ≥ 50 kg (110 lbs) and a body mass index ≥ 18 and ≤ 32 kg/m2
4. Women must be of non-childbearing potential:Surgically sterile; no menses for ≥ 12 months AND a follicle-stimulating hormone level>40 IU/L at screening; or meeting the definition of "postmenopausal range" based onscreening laboratory results
5. Willing and able to comply with all the study requirements and provide written informedconsent for the study

Exclusion Criteria:

1. Donated blood or experienced significant blood loss
2. Has inadequate venous access or unsuitable veins for venipuncture and IV administrationof the study drug
3. History of or have any evidence of diabetes mellitus
4. History of renal impairment or inflammatory bowel disease
5. History of clinically significant ear pathology, ear surgery, or hearing impairment
6. Active infection
7. History of malignancy
8. Have undergone a surgical procedure within 3 months prior to study entry or have anysurgical procedure anticipated to be required during the study.
9. Any clinically significant abnormality at screening that, inthe opinion of the Investigator, would exclude them from the study
10. Received the last dose of an investigational drug or treatment with a medical devicewithin 30 days or 5 half-lives prior to screening or currentlyparticipating in another study of an investigational drug or medical device
11. Previously participated in a study of IGF-1 or IGF-1R-related products
12. Any medical condition or laboratory abnormality, that in the opinion of the Investigator, would prevent the subject from completing the study, pose a risk to the subject, or confound the ability to interpret study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0 | during the study, up to 4 weeks

SECONDARY OUTCOMES:
ZB001 concentrations in the blood over time | Before and after drug administration, performed according to the protocol visit time specified in the plan. Up to 4 weeks
  PK parameters in the blood over time.
Serum ZB001 antidrug antibody (ADA) titers | Before and after drug administration, performed according to the protocol visit time specified in the plan. Up to 4 weeks
  antidrug antibody (ADA) titers of ZB001

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No